CLINICAL TRIAL: NCT04035590
Title: Seroma Reduction and Drain Free Mastectomy
Acronym: SARA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, James van Bastelaar, Surgeon, Principal Investigator, MD, PhD, Zuyderland Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METCZ2019016
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Seroma; Wound Complication
Keywords: Mastectomy; Drain
MeSH Terms: conditions — Breast Neoplasms; Seroma | interventions — Drainage

STUDY DESIGN:
Intervention Model Description: Study design is a randomized controlled trial. All patients are > 18 years and will be enrolled after obtaining informed consent in the surgical out patient clinics of Zuyderland Medical Center Sittard. All patients have an indication to undergo mastectomy due to invasive breast cancer or DCIS.
  Follow up will be performed until 6 months after surgery. Patients will be evaluated in the out patient clinic 1 week, 6 weeks, 3 months and 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With drain (Active Comparator): Patients undergo mastectomy with flap fixation and low vacuum drainage.
  Interventions: Procedure: With drain
- No drain (Experimental): Patients undergo mastectomy with flap fixation and low vacuum drainage is omitted.
  Interventions: Procedure: No drain

INTERVENTIONS:
Procedure: No drain — Mastectomy with flap fixation without low vacuum drainage
  Arms: No drain
Procedure: With drain — Mastectomy with flap fixation with low vacuum drainage
  Arms: With drain

SUMMARY:
To prove that omitting drains after mastectomy and flap fixation does not contribute to higher incidence of seroma formation and therefore reducing patient disutility such as seroma aspirations and visits to the outpatient clinic, as well as reducing seroma related wound complications.

DETAILED DESCRIPTION:
Rationale:

Seroma formation, a collection of serous fluid containing blood plasma and/or lymph fluid, is a common complication in breast cancer surgery and can lead to delayed wound healing, infection, skin flap necrosis, patient discomfort and repeated visits to the outpatient clinic and therefore extensive research has been done to further elucidate the pathophysiology and prevention of seroma formation. Promising results have resulted from studies focusing on flap fixation in order to reduce the incidence of seroma and seroma aspirations. Mastectomy with flap fixation is becoming standard practice and is currently combined with closed-suction drainage. Closed-suction drainage is considered gold standard for reducing seroma formation after breast cancer surgery. However, evidence shows that closed-suction drainage is insufficient in preventing seroma formation. One might wonder if there is still a place for closed-suction drainage after mastectomy if flap fixation is performed. The promising results in flap fixation could exclude drainage systems in breast cancer surgery. However, the available data consist of small case series and therefore a large randomized controlled trial is needed for it to be widely implemented.

To our knowledge, no randomized controlled trial has been conducted comparing flap fixation with and without closed-suction drainage with seroma aspiration as the primary outcome.

The investigators hypothesize that flap fixation with closed suction drainage does not cause a significant lower incidence of seroma aspirations, when compared to flap fixation alone. The investigators also expect that patients without drainage will experience significantly less discomfort and comparable rates of surgical site infections.

Objective: To prove that omitting drains after mastectomy and flap fixation does not contribute to higher incidence of seroma formation and therefore reducing patient disutility such as seroma aspirations and visits to the outpatient clinic, as well as reducing seroma related wound complications.

Study design: Prospective randomized controlled trial

Study population: Female patients > 18 years diagnosed with invasive breast cancer or DCIS (ductal carcinoma in situ) with an indication to perform mastectomy

Intervention (if applicable):

1. Mastectomy with flap fixation using sutures with closed suction drainage
2. Mastectomy with flap fixation using sutures without closed suction drainage

Main study parameters/endpoints:

Patients undergoing seroma aspiration (clinically significant seroma (CSS)).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients will be informed about the study before inclusion in the outpatient clinic. Informed consent will be obtained in the outpatient clinic a week after patients were initially informed. Postoperative check-ups will be done more frequently. Standard postoperative check-ups are planned at 2 weeks and 3 months. Additional study postoperative check-ups: 6 weeks, 6 months. Therefore, patients will be required to undergo two additional check-ups.

During out patients' visits, patients will hand in a questionnaire scale regarding cosmesis, pain and quality of life.

Patients will be clinically examined as they usually would be.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Female sex
* Indication for mastectomy

Exclusion Criteria:

* Patients undergoing breast conserving therapy
* Patients undergoing modified radical mastectomy
* Patients undergoing direct breast reconstruction
* Unable to comprehend implications and extent of study and sign for informed consent
* Patients with radiation therapy of unilateral breast in previous history

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 250 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Seroma aspiration of clinically significant seroma | During first six months post-operative
  Proportion of patients undergoing seroma aspiration of clinically significant seroma
  Clinically significant seroma defined as:
  1. Wound healing is at risk due to seroma (wound break down, seroma leakage, necrosis)
  2. There is discomfort or pain caused by large amounts of seroma, characterised by tenseness of the skin.
  3. There is contaminated/ infected seroma and aspiration is necessary to treat infection. All patients that undergo seroma aspiration due to infection will also be treated with a one week course of Augmentin 625 mg 3 times daily.

SECONDARY OUTCOMES:
Number of invasive interventions related to seroma or wound healing | During first six months post-operative
  Number of invasive interventions related to seroma or wound healing defined as: every aspiration of clinically significant seroma, incision and drainage of abscess or infected seroma and/or operative debriding of the wound.
Surgical site infection (SSI) rate | During the first six postoperative months
  Surgical site infection (SSI) rate, defined as redness, pain, heat or swelling at the site of the incision or by the drainage of pus. Infection rate will be measured by A) the need for antibiotics, B) seroma aspiration due to infection or C) surgical drainage.
Cosmesis | During the first six postoperative months
  Cosmesis rated by the patient using the numeric rating scale (NRS) every planned outpatient clinic visit.
Quality of life measured using the SF-12 Health Survey | During the first six postoperative months
  Quality of life measured using the SF-12 Health Survey. Resulting in 2 scores: the Mental Component Summary (MCS) and the Physical Component Summary (PCS). Both range between values of 0-100 with a score of 50 representing values of a standard population
The number of outpatient department visits | During the first six months postoperative.
  The number of outpatient department visits
Experienced pain: NRS | During the first six months postoperative
  Experienced wound pain and pain at the drain site by the patient using the NRS with a scale range from 0-10

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medisch Centrum, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Rooij L, van Kuijk SMJ, van Haaren ERM, Janssen A, Vissers YLJ, Beets GL, van Bastelaar J. A single-center, randomized, non-inferiority study evaluating seroma formation after mastectomy combined with flap fixation with or without suction drainage: protocol for the Seroma reduction and drAin fRee mAstectomy (SARA) trial. BMC Cancer. 2020 Aug 7;20(1):735. doi: 10.1186/s12885-020-07242-0. PMID 32767988